CLINICAL TRIAL: NCT03026842
Title: A Prospective, Randomized, Controlled Trial of Decitabine Versus Conventional Chemotherapy for Maintenance Therapy of Patients With Acute Myeloid Leukemia With t(8;21)
Brief Title: Decitabine Versus Conventional Chemotherapy for Maintenance Therapy of Acute Myeloid Leukemia With t(8;21)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The First Hospital of Jilin University (Other)
Collaborators: The Second Affiliated Hospital of Dalian Medical University (Other); Second Hospital of Jilin University (Other); Jilin University (Other)
Responsible Party: Principal Investigator, SuJun Gao, Head of Hematology Department, The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NECOG
Record Dates: First submitted 2017-01-15; First posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine; Daunorubicin; Cytarabine; NOAC protocol; aclacinomycins

ARMS (2):
- Decitabine (Experimental): Six cycles of decitabine IV over one hour at 20 mg/m2/day for 5 days, every 6 weeks
  Interventions: Drug: Decitabine
- Conventional chemotherapy (Active Comparator): Four cycles of conventional chemotherapy for 5 days, every 12 weeks. conventional chemotherapy includes in: DA regimen: Daunorubicin 45 mg/m2/day for 3 days, cytarabine 100 mg/m2/day for 5 days; MA regimen: Mitoxantrone 8 mg/m2/day for 3 days, cytarabine 100 mg/m2/day for 5 days; AA regimen: Aclacinomycin 20 mg/day for 5 days, cytarabine 100 mg/m2/day for 5 days.
  Interventions: Drug: Daunorubicin, Cytarabine; Drug: Mitoxantrone, Cytarabine; Drug: Aclacinomycin, Cytarabine

INTERVENTIONS:
Drug: Decitabine — 20 mg/m2/day for 5 days
  Arms: Decitabine
Drug: Daunorubicin, Cytarabine — Daunorubicin: 45 mg/m2/day for 3 days; Cytarabine: 100 mg/m2/day for 5 days
  Arms: Conventional chemotherapy
Drug: Mitoxantrone, Cytarabine — Mitoxantrone: 8 mg/m2/day for 3 days; Cytarabine: 100 mg/m2/day for 5 days
  Arms: Conventional chemotherapy
Drug: Aclacinomycin, Cytarabine — Aclacinomycin: 20 mg/day for 5 days; Cytarabine: 100 mg/m2/day for 5 days
  Arms: Conventional chemotherapy

SUMMARY:
Acute myeloid leukemia (AML) is the most common hematological malignancies in adult patients with leukemia, and t(8;21) AML accounts for a substantial proportion of AML. AML patients with t(8;21) possess a favorable outcome and 3 - 4 course high dose cytarabine (3 g/m2) is the standard consolidation therapy for these patients with a 5-year overall survival approximately 60%. In China, intermediate dose cytarabine (1 - 2 g/m2) is used for consolidation therapy due to toxicities. After 3 - 4 course cytarabine consolidation, maintenance therapy is performed with conventional chemotherapy with a 5-year overall survival approximately 60% as well. However, continuous chemotherapy may cause toxicities and inhibit patients' immune response. Exploring new drug for maintenance therapy is urgently needed. Decitabine has a potent ability to inhibit proliferation and induce apoptosis of AML1-ETO positive leukemia cell line. Furthermore, the immunomodulatory effect of decitabine was also reported by several studies. In this study, the investigators plan to carry out a prospective, multicenter, randomized, controlled trail to compare decitabine versus conventional chemotherapy for maintenance therapy of patients with AML with t(8;21). Results of this trial may optimize the treatment for AML patients with t(8;21) in the setting of intermediate dose cytarabine consolidation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are adults age ≥18 and ≤60 years
2. Patients are diagnosed as AML with t(8;21)
3. Continuous complete remission after induction and consolidation therapy with 3 - 4 course high dose cytarabine (2 g/m^2)
4. Patients whose aspartate transaminase (AST)/alanine transaminase (ALT) are ≤ 2.5 times higher than the normal upper limit, total bilirubin ≤ 3.0 mg/dl, and serum creatinine ≤ 2.0 mg/dl.
5. Subjects that signed the informed consent, which indicated they understood the purpose, the procedure and potential benefits of the trial and were willing to participate in the trial.

Exclusion Criteria:

1. Pregnant or lactating women.
2. ECOG performance status score > 2.
3. Patients are candidates for hematopoietic stem cell transplantation.
4. Patients with a history of use of azacitidine or decitabine.
5. Patients with mental or other disorders that cannot completely cooperate with the treatment or follow up.
6. Subjects that were allergic to decitabine vehicle.
7. Patients receive immunotherapy.
8. Patients also have other organ malignant tumor.
9. Participating in other clinical research in the same period.
10. The researchers estimate that patients cannot enter the clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-01; Primary Completion 2023-12 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Relapse free survival | Three years

SECONDARY OUTCOMES:
Overall survival | Three years
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From enrolling to two months after administrating the last course of decitabine or chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Su J Gao, PhD, Study Director — The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No